CLINICAL TRIAL: NCT01784744
Title: Hyperthermia and the Amelioration of Autism Symptoms
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Simons Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 12-10-113-01
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2014-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; ASD; Aspergers; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal samples collected for DNA and RNA extraction.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ASD Control: Patients aged 5 to 17 diagnosed with ASD.
  Interventions: Other: Hydroworx Pool at 102 degrees Fahrenheit
- ASD Case: Patients diagnosed with ASD aged 5 to 17 with a history of amelioration of symptoms during febrile episodes.
  Interventions: Other: Hydroworx Pool at 98 degrees Fahrenheit; Other: Hydroworx Pool at 102 degrees Fahrenheit

INTERVENTIONS:
Other: Hydroworx Pool at 98 degrees Fahrenheit
  Groups: ASD Case
Other: Hydroworx Pool at 102 degrees Fahrenheit

SUMMARY:
The febrile hypothesis of Autism Spectrum Disorder (ASD) stems from the observation that clinical symptoms improve during fever. This fever induced amelioration of symptoms could be due to one of three possible causes, (1) the direct effect of temperature; (2) a resulting change in the immune inflammatory system function associated with the infection or fever; and/or (3) and increase in the functionality of a previously dysfunctional Locus Coeruleus-Noradrenerigic (LC-NA) system. Little has been done to explore the potential direct effect an increased body temperature may have on autism symptomology. Parental reports have demonstrated that during febrile episodes children with ASD have improved social cognition and language skills, and decreased disruptive behaviors. In order to further explore the direct temperature effect, further investigation is needed, which the investigators propose below. The investigators propose to complete a one year double blind crossover study with 15 children with ASD between the ages of 5 and 17 years old. Five children with ASD will complete a control protocol prior to beginning the full protocol with 10 additional ASD children. This will allow for any needed amendment of protocol parameters prior to completion of the full protocol.

ELIGIBILITY:
ASD Controls Inclusion Criteria

* Aged 5 to 17
* Meets ASD criteria on the DSM-IV TR that is supported by the ADOS or the ADI-R

ASD Control Exclusion Criteria

* Children who are currently ill will not begin treatment until they are well.
* Females who are pregnant.
* Children who have abnormally high blood pressure prior to starting study treatment.
* Children with a BMI greater than 30.0 or below 18.5
* Children with history of seizures or cardiovascular problems

ASD Case Inclusion Criteria

* Meets ASD criteria on the DSM-IV TR that is supported by the ADOS or the ADI-R
* Aged 5 to 17
* Have a past history of improvement during febrile episodes

ASD Case Exclusion Criteria

* Children who are currently ill will not begin treatment until they are well.
* Females who are pregnant.
* Children who have abnormally high blood pressure prior to starting study treatment.
* Children with a BMI greater than 30.0 or below 18.5
* Children with history of seizures or cardiovascular problems

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 5 to 17 diagnosed with Autism Spectrum Disorder will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist | Screening, Day One and Day Two

SECONDARY OUTCOMES:
Social Responsiveness Scale | Screening, Day One, Day Two
Clinical Global Impression Scale - Improvement | Day One, Day Two

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York, United States